CLINICAL TRIAL: NCT06567314
Title: Phase 2 Study of Ivonescimab in Patients With Cutaneous Squamous Cell Carcinoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Summit Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-0501; NCI-2024-07130 (Other: NCI-CTRP Clinical Registry)
Record Dates: First submitted 2024-08-21; First posted 2024-08-22 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Cutaneous Squamous Cell Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Ivonescimab (Experimental): Participants found to be eligible to take part in this study, you will receive ivonescimab by vein over about 1-2 hours on Day 1 of each 21-day cycle (1 time every 3 weeks).
  Interventions: Drug: Ivonescimab

INTERVENTIONS:
Drug: Ivonescimab — Given by PO

SUMMARY:
To learn if ivonescimab can help to control advanced cSCC. The safety and effects of ivonescimab will also be studied.

DETAILED DESCRIPTION:
Primary Objective

- To determine the ORR of ivonescimab in patients with cSCC and CRPC

Secondary Objectives

* To evaluate other indicators of the antitumor efficacy of ivonescimab in patients with cSCC and CRPC.
* To evaluate the safety and tolerability of ivonescimab in patients with cSCC and CRPC

Exploratory Objective

* To evaluate potential predictors of response and resistance to ivonescimab
* To bank pre-treatment blood samples for future correlative analyses
* To evaluate imaging characteristics predictive of treatment response and side effects

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand and willingness to sign informed consent form prior to initiation of the study and any study procedures.
* Age ≥18 years.
* Has locally advanced surgically non-appropriate (unresectable and/or metastatic) cSCC (Cohort 1)..
* Has metastatic CRPC (Cohort 2):

  * Histologically or cytologically confirmed adenocarcinoma of the prostate without neuroendocrine differentiation or small cell histology.
  * Documented prostate cancer progression as documented by PSA progression according to PCWG3 criteria.
  * Surgically or medically castrated, with serum testosterone level <50 ng/dL.
* Refractory or naïve to anti-PD-1 therapy (Cohort 1). There is no limit on the number of prior lines of therapy. NOTE: Detailed information regarding duration of prior anti-PD-1 therapy and the extent of progression at the time of anti-PD-1 therapy discontinuation will be collected.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 (Appendix 1).
* Cohort 1: measurable disease per the RECIST v1.1 or Measurable by mRECIST for skin cancer or Global Assessment or Papillary/Ulceration Response Assessment or Pathological Assessment or WHO Criteria for Response Assessment in Cutaneous Squamous Cell Carcinoma, as appropriate (Appendix 4).
* Adequate organ and marrow function as defined below within 28 days of study treatment initiation:

  * Hemoglobin >9.0 g/dL
  * Absolute neutrophil count ≥1500/mL
  * Platelets ≥100,000/mL
  * Total bilirubin ≤1.5 institutional upper limit of normal (ULN). Documented Gilbert syndrome is allowed if total bilirubin is ≤3 × ULN.
  * AST/alanine transaminase ≤2.5 × institutional ULN. Transaminases up to 3 × ULN in the presence of liver metastases.
  * Serum creatinine ≤1.5 × ULN OR measured or calculated creatinine clearance (CrCl; glomerular filtration rate can also be used in place of creatinine or CrCl) ≥60 mL/min for participants with creatinine levels >1.5 × institutional ULN (CrCl should be calculated per institutional standard).
  * Urine protein <2+ or 24-hour urine protein quantification <1.0 g
  * For participants not receiving therapeutic anticoagulation: international normalized ratio or activated partial thromboplastin time ≤1.5 × ULN. For patients receiving therapeutic anticoagulation: stable anticoagulant regimen.
  * Albumin >2.5 mg/dL.
* Participants must have adequate washout from prior therapy at the time of study treatment initiation: 4 weeks from major surgery; 4 weeks from antibody-based therapy; 2 weeks or 5 half-lives (whichever is shorter) from any targeted therapy or small molecule therapy; 3 weeks or 5 half-lives (whichever is shorter) from chemotherapy or 6 weeks in the case of certain therapies (e.g., extensive radiotherapy, mitomycin C, and nitrosoureas); 4 weeks from radiation therapy; and at least 2 weeks from palliative radiotherapy.
* Prior treatment with anti-VEGF therapy is allowed (Cohort 1).
* Adequately controlled blood pressure with 0 or 1 antihypertensive medication (defined as blood pressure ≤150/100 mmHg at screening and no changes in antihypertensive medication within 7 days of Day 1 Cycle 1.
* Women of childbearing potential (WOCBP) should have a negative urine or serum pregnancy within 72 hours prior to study treatment initiation. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
* WOCBP must agree to use adequate contraception during the study treatment period and for 120 days after completion of study treatment. A woman is considered to be of childbearing potential if she is postmenarcheal, has not reached a postmenopausal state (≥12 continuous months of amenorrhea with no identified cause other than menopause), and is not permanently infertile due to surgery (i.e., removal of ovaries, fallopian tubes, and/or uterus) or another cause as determined by the investigator (e.g., Müllerian agenesis). Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.
* Male participants of childbearing potential must agree to use adequate contraception during the study treatment period and for 120 days after completion of study treatment.

Exclusion Criteria:

* Patients who have previously been treated with PD-1/PD-L1 inhibitors and required permanent discontinuation, or systemic immunosuppression due to irAEs.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to ivonescimab.
* Pregnant or breastfeeding.
* Participants with an active, known or suspected autoimmune disease. Participants with type I diabetes mellitus, hypothyroidism only requiring hormone replacement, skin disorders (such as vitiligo, psoriasis, or alopecia) not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are permitted to enroll.
* Known history of positive test for human immunodeficiency virus or known acquired immunodeficiency syndrome.
* Known history of acute or chronic hepatitis B virus or hepatitis C virus infection.
* Previous solid organ or allogeneic hematopoietic stem cell transplant.
* Active infection requiring IV antibiotics or other uncontrolled intercurrent illness requiring hospitalization.
* Unresolved toxicities from prior therapy (defined as having not resolved to NCI CTCAE v.5.0 Grade ≤1 or baseline) or any other toxicity that is deemed irreversible by the investigator. Exceptions include endocrinopathies from prior therapy or disease and successfully treated (such as hypothyroidism, diabetes mellitus), alopecia, vitiligo, and Grade ≤2 peripheral neuropathy.
* Major blood vessel invasion.
* Major surgical procedures or serious trauma within 4 weeks prior to study treatment initiation, or plans for major surgical procedures within 4 weeks after the first dose of study treatment (as determined by the investigator). Minor local procedures (excluding central venous catheterization and port implantation) within 3 days prior to study treatment initiation.
* Unstable angina, myocardial infarction, congestive heart failure (New York Heart Association [NYHA] classification Grade ≥2) or vascular disease (e.g., aortic aneurysm at risk of rupture) that required hospitalization within 12 months prior to study treatment initiation, or other cardiac impairment that may affect the safety evaluation of the study drug (e.g., poorly controlled arrhythmias, myocardial ischemia).
* History of esophageal gastric varices, severe ulcers, wounds that do not heal, abdominal fistula, intra-abdominal abscesses, or acute gastrointestinal bleeding within 6 months prior to study treatment initiation.
* History of arterial thromboembolic event, venous thromboembolic event of Grade ≥3 as specified in NCI CTCAE v5.0, transient ischemic attack, cerebrovascular accident, hypertensive crisis, or hypertensive encephalopathy within 6 months prior to study treatment initiation.
* Acute exacerbation of chronic obstructive pulmonary disease within 4 weeks prior to study treatment initiation.
* History of perforation of the gastrointestinal tract and/or fistula, history of gastrointestinal obstruction (including incomplete intestinal obstruction requiring parenteral nutrition), extensive bowel resection (partial colectomy or extensive small bowel resection) within 6 months prior to study treatment initiation.
* Treatment with a live, attenuated vaccine within 4 weeks prior to study treatment initiation, or anticipation of need for such a vaccine during the course of the study.
* Has a known additional malignancy that is progressing or requires active treatment.

Exceptions include basal cell carcinoma of the skin, squamous cell carcinoma of the skin that has undergone potentially curative therapy, or in situ cervical cancer.

* Has a known psychiatric or substance abuse disorder that would interfere with cooperation with the requirements of the study.
* Inability to comply with the study and follow-up procedures.
* Participants who are receiving any other investigational agents.
* Participants with psychiatric illness/social situations that would limit compliance with study requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-12-02 (Actual); Primary Completion 2028-09-01 (Estimated); Study Completion 2030-09-01 (Estimated)

PRIMARY OUTCOMES:
Safety and adverse events (AEs) | Through study completion; an average of 1 year.
  Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Aung Naing, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org